CLINICAL TRIAL: NCT01356420
Title: Smith-Lemli-Opitz Syndrome: A Longitudinal Clinical Study of Patients Receiving Cholesterol Supplementation
Brief Title: Sterol and Isoprenoid Disease Research Consortium: Smith-Lemli-Opitz Syndrome
Acronym: STAIR-SLOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: NICHD cut funding
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jean-Baptiste Roullet, Clinical Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAIR 7001
Record Dates: First submitted 2011-05-11; First posted 2011-05-19 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: SLOS
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cholesterol supplementation (Experimental): All new subjects will come to their first visit with an least 3 weeks of stable cholesterol intake. Typically and preferably this will include egg yolk as cholesterol supplement, but in some instances e.g. intolerance to egg yolk it may include a new encapsulated cholesterol preparation, Sloesterol.
  Interventions: Dietary Supplement: Cholesterol supplementation

INTERVENTIONS:
Dietary Supplement: Cholesterol supplementation — Cholesterol supplementation may be achieved with SLOesterol instead of or in combination with egg yolk. SLOesterol is a powder formulation that contains cholesterol and natural emulsifier. It is considered a medical food developed by Solace Nutrition and available by prescription only.

SUMMARY:
The purpose of this study is to learn about Smith-Lemli-Opitz Syndrome (SLOS). SLOS is an inherited condition that is caused by the body not making an enzyme as it should. The body needs the enzyme to help make cholesterol. SLOS can cause many health problems including slow growth and development, eating disorders, sleep disorders, behavior disorders, and eye diseases. Severe SLOS leads to birth defects and mental retardation and in many cases early death. The investigators plan to measure cholesterol and other sterol levels, perform clinical observations, whole body testing and imaging (brain MRIs), to learn more about the disease and its progression, differences in the clinical features among individuals with SLOS, and look at the effect of cholesterol supplementation in this condition.

The study is an interventional study to characterize disease progression and correlations between clinical, biochemical and physiological features of the disease. The main hypothesis is that dietary cholesterol supplementation does not improve features of SLOS related to the brain (e.g. IQ, behavior).

DETAILED DESCRIPTION:
Smith-Lemli-Opitz syndrome (SLOS) is a disorder of cholesterol synthesis, or production. It is caused by mutations in the DHCR7 gene which encodes for 7-dehydrocholesterol- Δ7-reductase, an enzyme necessary for the production of cholesterol in the body. Affected individuals exhibit multiple malformations and mental retardation. The features of SLOS are thought to be primarily related to cholesterol deficiency and accumulation of cholesterol precursors. However, the clinical phenotype is not well characterized, the biochemical pathogenesis is incompletely understood, and there is no proven therapy for this devastating condition. Thus our primary objective is to better define the clinical and biochemical phenotypes of the disease using a natural history study design. The study will contribute to creating a comprehensive SLOS patient registry, identify biomarkers that can be used for diagnostic testing, screening and outcome measures in future therapeutic trials. All patients with SLOS receive dietary cholesterol supplementation with the hope that cholesterol supplementation will improve the clinical manifestation of the disease. However, there is no evidence supporting a clinical benefit of cholesterol supplementation. Thus a secondary objective of the study is to determine if cholesterol intake correlates with changes in whole body cholesterol homeostasis and clinical end-points.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Smith-Lemli-Opitz Syndrome (SLOS)
* Males and females of all ages
* Willing and able to travel to OHSU or another STAIR site

Exclusion Criteria:

* Subject does not have Smith-Lemli-Opitz Syndrome (SLOS)

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To define the rate of progression of clinical and biochemical measures in patients with Smith Lemli-Opitz syndrome receiving dietary cholesterol supplementation. | Once per year at annual study visit
  This study will measure changes in whole body cholesterol pool size, 24S, cholesterol absorption and synthesis in relation with cholesterol intake and changes in clincal end-points.

SECONDARY OUTCOMES:
Correlate biochemical and clinical phenotypes | Once per year at annual study visit
  To correlate biochemical and clinical phenotypes in SLOS subjects given dietary cholesterol with changes in whole body cholesterol pool size, and with its major determinants (cholesterol synthesis, absorption and intake).
Identify clinical or biochemical markers for future therapeutic trials. | Once per year at annual study visit
  To identify clinical or biochemical markers that can be used as outcome measures in a future therapeutic trial.
Identify a biochemical marker that can be used for diagnostic testing or screening. | Once per year at annual study visit
  To identify a biochemical marker that can be used for diagnostic testing or screening
Develop a registry and repository of biomaterials of SLOS patients | each subject will be enrolled in the registry at the baseline/initial visit, if they choose to participate in this portion of the study
  To develop a registry of well characterized SLOS patients and to maintain a repository of biomaterials corresponding to these patients

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steiner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - Pdgen, Nichd, Nih, Dhhs, Bethesda, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children'S Hospital of Pittsburgh of Upmc, Pittsburgh, Pennsylvania